CLINICAL TRIAL: NCT05859672
Title: A Study of Intraoperative Transpulmonary and Intrathoracic Pressure Changes Associated With Ventilator Management of Tidal Volume and Positive End-expiratory Pressure (PEEP)
Brief Title: Ventilation and Esophageal Pressure Changes
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1903822
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study to observe the effect of variations in ventilator settings including tidal volume and PEEP on transpulmonary pressure monitored with an esophageal balloon catheter and to correlate intraoperative transpulmonary pressure variations and intraoperative stroke volume variation changes.

DETAILED DESCRIPTION:
This study seeks to observe the effects of variations in ventilator settings on transpulmonary and intrathoracic pressures. More specifically, to observe the impact of variations in tidal volume from 6 mL/kg to 8 mL/kg and PEEP from 0 cm of water (H2O) to 5 cm H2O on transpulmonary and intrathoracic pressures monitored with an esophageal balloon catheter. The impact of this recommended decrease in tidal volume on the clinical utility of stroke volume variation (SVV) as a guide for fluid administration has not been previously examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery requiring general anesthesia and endotracheal intubation.
* Age ≥ 18

Exclusion Criteria:

* Patients undergoing planned esophageal surgery
* Patients with significant nasal or esophageal pathology
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Intrathoracic Pressure | Intra-operative
  Measure the intrathoracic pressure changes monitored with an esophageal pressure balloon catheter associated with intraoperative changes in mechanical ventilation parameters such as tidal volume and PEEP

SECONDARY OUTCOMES:
Stroke Volume Variation | Intra-operative
  Characterizing the changes in SVV associated with intraoperative changes in mechanical ventilation parameters such as tidal volume and PEEP and the correlations with changes in intrathoracic pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States